CLINICAL TRIAL: NCT06076473
Title: Pilot Untargeted Metabolomics for Primary Aldosteronism in Plasma (PUMPAP)
Brief Title: Untargeted Metabolomics for Primary Aldosteronism
Acronym: PUMPAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: LHS001
Record Dates: First submitted 2022-12-30; First posted 2023-10-10 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-12

CONDITIONS: Primary Aldosteronism
Keywords: Pilot; Untargeted Metabolomics; Primary Aldosteronism; Plasma
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Surplus lithium heparin samples collected as part of routine care will be stored prior to analysis and used to destruction during analysis. Spare aliquots for data validation will be stored until the end of the study period (2 years) and then discarded in line with standard laboratory protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Confirmed Primary Aldosteronism: Confirmed Primary Aldosteronism
  Interventions: Diagnostic Test: Untargeted metabolomics
- Non-Primary Aldosteronism: Other causes of hypertension
  Interventions: Diagnostic Test: Untargeted metabolomics

INTERVENTIONS:
Diagnostic Test: Untargeted metabolomics — Pilot untargeted plasma metabolomics aiming to identify novel biomarkers for PA diagnosis and subtyping, which could be compared against existing biomarkers and taken forward to larger future studies.

SUMMARY:
Primary aldosteronism (PA) is a common and likely under-diagnosed cause of secondary hypertension with associated cardiovascular morbidity and mortality. Current diagnosis comprises screening, confirmatory testing and sub-type classification (lateralisation) to distinguish unilateral disease (requiring surgery) from bilateral disease (requiring medical management). This multi-step process is complex and variable with a lack of uniformity in diagnostic protocols, standardised/reference assay methodologies, and diagnostic thresholds. There is evidence in the literature that targeted serum steroid panels may have a role in diagnosis of PA, and both targeted steroid panels and untargeted metabolomics in serum and urine are a promising area of research.

This study aims to identify and recruit participants (n=40; 20 with confirmed PA and 20 with other causes of hypertension) willing to donate lithium heparin plasma for a metabolomics pilot study. This plasma will be interrogated through untargeted metabolomics using gas/liquid chromatography-mass-spectrometric methods and computational data processing to allow power calculations and inform experimental design for future studies. The utility of metabolites from the metabolomics dataset will be evaluated by comparison against current biomarkers for screening, diagnosis and lateralisation as well as radiology and histology acquired through routine diagnostic work-up. The long-term aim for larger studies is to identify suitable candidate analytes in plasma for future development into targeted, clinically-useful analyte panels.

DETAILED DESCRIPTION:
Participant Recruitment

* Suitable participants will be identified by members of their care teams, for whom screening, confirmatory testing and lateralisation will be / have been completed at LUHFT.
* Potential participants will be approached by a member of the study team seeking consent. Saline infusion testing and adrenal vein sampling are key points in the diagnostic work-up for participant recruitment for non-PA and PA cohorts, respectively.
* Consenting participants will have lithium heparin plasma collected and stored until the requisite sample size has been reached (n=40; 20 with PA and 20 with PA excluded by aldosterone:renin ratio at screening or saline infusion confirmatory testing). A lithium heparin tube will be used for routine renal profiles requested as part of saline infusion tests or adrenal vein sampling to avoid requirements for any additional blood tubes. The sample will be centrifuged and separated into two aliquots. One aliquot for metabolomic analysis at the University of Liverpool and one for storage within LUHFT until the end of the study (2 years) in case data validation is required. Clinical, biochemical, radiological and histological information from routine care will help to classify participants into PA (n=20) and non-PA (n=20) groups, as well as to assign lateralisation status. Ideally there will be equal representation from unilateral left, unilateral right and bilateral disease in the PA sub-set.
* Recruitment will close after 18 months.

Laboratory Analysis

* Untargeted metabolomics analysis using chromatography-mass spectrometric methods will be performed on lithium heparin plasma from all consenting participants. An aliquot of this sample will be transferred to the University of Liverpool for analysis and used to destruction (with no backwards transfer).

Data Analysis

* Computation analysis of the data set will be used to screen for novel PA biomarkers that could be further investigated in later studies.
* Univariate and multivariate methods will be applied. These will include univariate statistical and AUROC calculations, adjusted logistic regression techniques, unsupervised (clustering/visualisation) and supervised (classifier-based) multivariate methods
* Power calculations and pilot data set analysis will inform future experimental design.

Sample Storage

* Primary aliquots will be stored at LUHFT for up to 18 months awaiting analysis. They will then be transferred in one batch to the University of Liverpool and used to destruction.
* Secondary aliquots of biological material (which are intended as a back-up in case data validation is required) will be stored under appropriate conditions to preserve integrity until the end of the study. Samples will be disposed of after completion of the pilot study (2 years) in line with routine laboratory practice.

Data storage

* Storage of analytical and metadata will be for a period of five years. It will be stored on a secure computer on the Royal Liverpool University Hospital (RLUH) network.

ELIGIBILITY:
Inclusion Criteria:

Screening for PA to be performed in people with:

* sustained blood pressure (BP) above 150/100 mm Hg on each of three measurements obtained on different days, with hypertension (BP >140/90 mm Hg) resistant to three conventional antihypertensive drugs (including a diuretic), or controlled BP (<140/90 mm Hg) on four or more antihypertensive drugs.
* hypertension and spontaneous or diuretic-induced hypokalaemia.
* hypertension and adrenal incidentaloma.
* hypertension and sleep apnoea.
* hypertension and a family history of early onset hypertension or cerebrovascular accident at a young age (<40 years).
* all hypertensive first-degree relatives of people with PA.

Subset of people being screened for PA who are eligible for inclusion in this study:

* 18 years of age or older.
* People under the care of LUHFT.
* Able to give informed consent.
* Having lithium heparin plasma samples collected as part of their routine care.

Exclusion Criteria:

* Under 18 years of age.
* Unable to give informed consent.
* Insufficient clinical/biochemical/radiological/histological information to accurately assign patients to PA or non-PA subsets.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be undergoing diagnostic work-up for PA, meet the above eligibility criteria, and give informed consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2025-01-19 (Estimated); Study Completion 2025-01-19 (Estimated)

PRIMARY OUTCOMES:
Untargeted metabolomics | 2 years
  Identification of candidate biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Davies, MChem MSc, Principal Investigator — Liverpool University Hospitals NHS Foundation Trust
Locations (1):
- Liverpool University Hospitals NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Patient identifiable data will not be shared outside the study team. Data will be pseudo-anonymised (mapped onto a unique study ID) by the study team to remove direct traceability to the participant and allow data to be shared between participating sites.